CLINICAL TRIAL: NCT05926934
Title: A Single-center, 3-arm, Parallel-group Randomized Controlled Trial to Evaluate Bond Failures and the Effectiveness of Three Orthodontic Retention Schemes in Preventing Post-treatment Mandibular Arch Changes
Brief Title: The Effectiveness of 3 Orthodontic Fixed Retention Schemes on Post-treatment Stability and Gingival Recession
Acronym: OrthRe10tion
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Iosif Sifakakis, Associate Professor, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 409/08.02.2022
Record Dates: First submitted 2023-05-31; First posted 2023-07-03 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Relapse; Orthodontic Retention
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Single strand β-Ti fixed retainer (Experimental): Single strand β-Ti fixed retainer 0.011in diameter, bonded on each tooth separately from #33-43
  Interventions: Device: Experimental: Single strand β-Ti fixed retainer
- SS fixed retainer (Experimental): SS fixed retainer 0.028in diameter, bonded on each tooth separately from #33-43
  Interventions: Device: Experimental: SS fixed retainer
- Twisted fixed retainer (Experimental): Twisted fixed retainer 0.027in diameter, bonded on each tooth separately from #33-43
  Interventions: Device: Experimental: Twisted fixed retainer

INTERVENTIONS:
Device: Experimental: Single strand β-Ti fixed retainer — All 90 patients between 13-30 y.o. treated with fixed orthodontic appliances (Roth 0.018'' slot at their final finishing stage) on at least between their lower first premolars and with no lower anterior teeth crowding (total irregularity index score = 0) and no need of removable retention appliances on their lower teeth, were randomly assigned to one of the three experimental groups.
  Arms: Single strand β-Ti fixed retainer
Device: Experimental: SS fixed retainer — All 90 patients between 13-30 y.o. treated with fixed orthodontic appliances (Roth 0.018'' slot at their final finishing stage) on at least between their lower first premolars and with no lower anterior teeth crowding (total irregularity index score = 0) and no need of removable retention appliances on their lower teeth, were randomly assigned to one of the three experimental groups.
  Arms: SS fixed retainer
Device: Experimental: Twisted fixed retainer — All 90 patients between 13-30 y.o. treated with fixed orthodontic appliances (Roth 0.018'' slot at their final finishing stage) on at least between their lower first premolars and with no lower anterior teeth crowding (total irregularity index score = 0) and no need of removable retention appliances on their lower teeth, were randomly assigned to one of the three experimental groups.
  Arms: Twisted fixed retainer

SUMMARY:
There is high possibility of relapse of the lower anterior teeth after orthodontic treatment. Relapse is related with the initial orthodontic anomaly, pathology of surrounding tissues, patient's age and sex and compliance and the retention protocol applied. The options for the later are various. Permanent fixed retainers are considered of the most common ones and vastly vary based of composition. There are fixed retainers distinguished for their composition (SS, β-NiTi, fiber-reinforced composite retainers) or for their shape and dimensions (round or rectangular shape and single-strand or multi-strand respectively), and/or for the teeth they are placed on (canine and canine or canine to canine). Fixed retainers may require patient's cooperation , nevertheless debond failure rate varies between 0.1-53%.

The aim of this prospective randomized clinical study is to compare failure incidents and retention effect on lower anterior teeth after orthodontic finish between three different types of fixed retainers. There will be 3 arms studied in this research: a) single strand 0.016x0.022'' β-Ti canine to canine, b) 0.028'' SS canine to canine and c) 0.027'' multi-strand twistflex canine to canine. Variables such as repeatability of failures, and undesired tooth movements will be measured. Measurements will be repeated every 3 months after patient's recruitment in this study, for one year period (12 months in total). Intraoral scans will be collected during baseline (fixed retainer insertion) and after 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with fixed orthodontic appliances (Roth 0.018'' slot at their final finishing stage)
* Patients with fixed orthodontic appliances at least between their lower first premolars
* No lower anterior teeth crowding (total irregularity index score = 0)
* Patients with no need of removable retention appliances on their lower teeth

Exclusion Criteria:

* Active caries on adjacent or lingual surfaces of lower anterior teeth
* Active periodontitis
* Supragingival calculus
* Gum bleeding during bonding of fixed retainer
* Gingival pocket depth greater than 3mm
* Syndromes or other anomalies of the craniofacial complex or other mental illness
* Missing or impacted teeth or other dental anomalies
* Congenital anomalies/syndromes
* Allergies regarding the alloys of fixed retainers
* Need for chemoprevention before data collection of periodontal indexes
* Diabetes
* Smoking
* Usage of antibiotics
* Pregnancy
* Participation in other clinical trials

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-01-16 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Number of teeth that failed regarding the bonding strength | baseline-3 months
Number of teeth that failed regarding the bonding strength | 3 months-6 months
Number of teeth that failed regarding the bonding strength | 6 months-9 months
Number of teeth that failed regarding the bonding strength | 9 months-1 year
Repeatability of bonding strength failure per patient and per tooth | baseline-3 months
Repeatability of bonding strength failure per patient and per tooth | 3 months-6 months
Repeatability of bonding strength failure per patient and per tooth | 6 months-9months
Repeatability of bonding strength failure per patient and per tooth | 9months-1 year
Breakage of fixed retainer wires | baseline-3 months
Breakage of fixed retainer wires | 3 months-6 months
Breakage of fixed retainer wires | 6 months-9 months
Breakage of fixed retainer wires | 9 months-1 year
Space discrepancy (Little index)(in mm) | baseline-3 months
Space discrepancy (Little index)(in mm) | 3 months-6 months
Space discrepancy (Little index)(in mm) | 6 months-9 months
Space discrepancy (Little index)(in mm) | 9 months-1 year
Mandibular intercanine distance | baseline-3 months
Mandibular intercanine distance | 3 months-6 months
Mandibular intercanine distance | 6 months-9 months
Mandibular arch length (in mm) | 9 months-1 year

SECONDARY OUTCOMES:
Tooth rotations in lower anterior teeth | baseline-3 months
Tooth rotations in lower anterior teeth | 3 months-6 months
Tooth rotations in lower anterior teeth | 6 months-9 months
Tooth rotations in lower anterior teeth | 9 months-1 year
Extrusion in lower anterior teeth | baseline-3 months
Extrusion in lower anterior teeth | 3 months-6 months
Extrusion in lower anterior teeth | 6 months-9 months
Extrusion in lower anterior teeth | 9 months-1 year
Tip inclinations anteroposteriorly | baseline-3 months
Tip inclinations anteroposteriorly | 3 months-6 months
Tip inclinations anteroposteriorly | 6 months-9 months
Tip inclinations anteroposteriorly | 9 months -1 year

CONTACTS AND LOCATIONS:
Locations (1):
- National and Kapodistrian University of Athens, School of Dentistry, Departments of Orthodontics, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No